CLINICAL TRIAL: NCT00810329
Title: Identify Unique Set of Proteins in Cerebrospinal Fluid, Which Are Believed to be Found in Chronic Fatigue Syndrome Participants, But Not in Healthy Controls.
Brief Title: Proteomics of Cerebrospinal Fluid in Chronic Fatigue Syndrome
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); University of South Alabama (Other)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Other Study IDs: 2006-481; R01ES015382 (NIH)
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Fatigue Syndrome; Fibromyalgia; Gulf War Illness; Multiple Chemical Sensitivity; Interstitial Cystitis; Irritable Bowel Syndrome
Keywords: CFS,FM,CSF,Proteomics,Pain,Fatigue,GWI,IBS,IC,MCS.
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fibromyalgia; Multiple Chemical Sensitivity; Cystitis, Interstitial; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cheek swabs, on the right and left inner cheek. Others:Cerebrospinal fluid samples,Blood samples Urine samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: This group consists of patients with Chronic fatigue syndrome, Fibromyalgia and other conditions like Multiple chemical sensitivity, Irritable bowel syndrome, Interstitial Cystitis, Gulf War Illness.
- 2: The healthy control group

SUMMARY:
The purpose of this study is:

1. To identify specific set of proteins in the cerebrospinal fluid (fluid surrounding the brain and the spinal cord), that are believed to be seen in Chronic fatigue syndrome (CFS) patients, but not in healthy controls (HC). A similar study that the investigators had conducted before,suggested that significant changes in proteins in the cerebrospinal fluid may be due to the fundamental pathology of this disorder.
2. Increased cerebrospinal fluid pressure (pressure that helps the cerebrospinal fluid to move around the brain and the spinal cord), may be related with certain symptoms like headache, sleep problems, light headedness, increased pain, excessive tiredness (fatigue) even with minimal work and memory problems.
3. Assessment of Autonomic Nervous system function (Sympathetic nervous system)between the CFS and HC.
4. Perform Lung Function Testing or pulmonary function test to estimate the lung capacities and score shortness of breath while performing breathing maneuvers.
5. Dolorimetry (18 tender point test) for assessment of pain threshold.
6. Capsaicin skin test
7. Allergy skin test

DETAILED DESCRIPTION:
Neurological dysfunction is a key component of the clinical expression and case designation of chronic fatigue syndrome (CFS), fibromyalgia (FM)and other related conditions.If the central nervous system is involved, then evidence will be present in the cerebrospinal fluid. Distinct patterns of proteins will be present in Chronic fatigue syndrome (CFS) compared to healthy control (HC) subjects.

Other testing in our study would include:

1. a)Assessment of lung function and capacities. Additional interests are to assess the shortness of breath, lightheadedness, headache and chest tightness during the breathing maneuvers. The rationale for recording these symptoms is to understand the pathophysiology of sensory disturbances that are more noted in the CFS and Fibromyalgia group, but not in HC.
2. Compare the blood pressure and heart rate response before and after hand grip exercise testing. This is a test to measure the Autonomic Nervous system function (Sympathetic nervous system).
3. Skin tests like:

   i) Capsaicin skin test, to check for specific responses like burning sensation, area of skin redness, itchy sensation to varying doses of capsaicin (essence of chilli pepper), when placed on the forearm and to compare if there are any differences seen between the responses in CFS and Healthy controls.

   ii) Allergy skin test to look if there are any allergies that are seen in the set of CFS population.
4. 18 tenderness point testing to compare the pain threshold before and after the lumbar puncture also know as the spinal tap. 18 tenderness point testing is a diagnostic test for Fibromyalgia.
5. Many of the participants with CFS do have associated Migraine headaches and they complain of severe light and sound sensitivity. We are analysing those group of people and decision have to be made as to which medications would work at best, thus providing immediate relief from headache.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic Fatigue Syndrome
2. Fibromyalgia
3. Gulf War Illness
4. Multiple Chemical Sensitivity
5. Irritable Bowel Syndrome
6. Interstitial Cystitis

Exclusion Criteria:

1. You do not want to have a lumbar puncture performed.
2. You have a severe physical impairment that does not permit lumbar puncture or completion of the remainder of the tests (e.g. severe scoliosis or curvature of the back).
3. You have a medical condition with symptoms similar to Chronic Fatigue Syndrome such as regional pain syndromes, reflex sympathetic dystrophy, morbid obesity, autoimmune / inflammatory diseases, cardiopulmonary disorders), neurological disorders (e.g. seizures, dementia, degenerative disorders), uncontrolled endocrine or allergic diseases or, cancer.
4. You have a severe psychiatric illness such as schizophrenia, substance abuse, major depression with previous suicidal attempts, gestures or ideas about committing suicide.
5. You are mentally retarded or cannot understand this informed consent, cannot provide absolute willingness to have a lumbar puncture as part of this study, or are unable to complete the questionnaires and other studies that are part of this research project
6. You are in jail or prison.
7. You are pregnant.
8. You smoke more than 5 cigarettes per day. You will be allowed to taper your smoking before your participation in the actual study visit. This is an excellent opportunity to ask about our Smoking Cessation Programs.
9. You drink or eat caffeine containing products with more than the equivalent of 2 cups of coffee. You will be allowed to taper your caffeine intake before the study visit.
10. You have used narcotics or other illegal medications for more than 3 months. These will be discussed with Dr. Baraniuk.
11. You have a positive HIV test, or blood, liver or kidney tests that are abnormal.
12. You are participating only so you can be paid for taking part in this spinal tap study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Georgetown University Division of Rheumatology, Immunology and Allergy and other Divisions
  2. IRB-approved websites and support groups.
  3. IRB- approved advertisments
  4. Self-referral.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2007-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Differences in the proteins in the fluid around the brain, between Chronic fatigue syndrome and Healthy subjects. These proteins may identify the disease and define its mechanism. | 3 - 4 years

SECONDARY OUTCOMES:
Blood pressure differences in response to exercise, blood test and cerebrospinal fluid, questionnaire results and sensory nerve testing to determine the role(s) of altered nerve and brain function in Chronic fatigue syndrome. | 3- 4 years

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, MD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, 3800 Reservoir Rd NW, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Baraniuk JN, Casado B, Maibach H, Clauw DJ, Pannell LK, Hess S S. A Chronic Fatigue Syndrome - related proteome in human cerebrospinal fluid. BMC Neurol. 2005 Dec 1;5:22. doi: 10.1186/1471-2377-5-22. PMID 16321154
- [Derived] Ravindran MK, Zheng Y, Timbol C, Merck SJ, Baraniuk JN. Migraine headaches in chronic fatigue syndrome (CFS): comparison of two prospective cross-sectional studies. BMC Neurol. 2011 Mar 5;11:30. doi: 10.1186/1471-2377-11-30. PMID 21375763
- See also: Laboratory Website — http://www9.georgetown.edu/faculty/baraniuj/Site/Current_Research.html